CLINICAL TRIAL: NCT02052726
Title: A Phase 1, Placebo-controlled, Randomized, Observer-blinded Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of An Adjuvanted Clostridium Difficile Vaccine Administered As A 3-dose Regimen In Healthy Adults Aged 50 To 85 Years
Brief Title: A Study To Investigate A Clostridium Difficile Vaccine In Healthy Adults Aged 50 To 85 Years, Who Will Each Receive 3 Doses Of Vaccine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Prevention
Other Study IDs: B5091002
Record Dates: First submitted 2013-12-17; First posted 2014-02-03 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Clostridium Difficile
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm Label: Month 0, 1 and 3 Schedule (Experimental)
  Interventions: Biological: C. difficile vaccine with adjuvant; Biological: Placebo
- Day 1, 8, and 30 Schedule (Experimental)
  Interventions: Biological: C. difficile vaccine with adjuvant; Biological: placebo

INTERVENTIONS:
Biological: C. difficile vaccine with adjuvant — C. difficile vaccine with adjuvant administered at Month 0, 1, and 3.
  Arms: Arm Label: Month 0, 1 and 3 Schedule
Biological: Placebo — Placebo administered at Month 0, 1, and 3.
  Arms: Arm Label: Month 0, 1 and 3 Schedule
Biological: C. difficile vaccine with adjuvant — C. difficile vaccine with adjuvant administered at day 1, 8, 30.
  Arms: Day 1, 8, and 30 Schedule
Biological: placebo — Placebo administered at Day 1, 8, and 30.
  Arms: Day 1, 8, and 30 Schedule

SUMMARY:
This study will investigate a clostridium difficile vaccine in healthy adults aged 50 to 85 years, who will each receive 3 doses of vaccine. Subjects will receive their vaccine doses at either months 0, 1, and 3 or days 1, 8, and 30. Subjects will be divided into 2 age groups (50-64 and 65-85 years of age). The study will assess how safe and tolerable the vaccine is, and also look at subjects' immune response to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults aged 50 to 85 years at enrollment

Exclusion Criteria:

* Proven or suspected prior episode of Clostridium difficile associated diarrhea.
* Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 8 weeks before receipt of study vaccine.
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2015-05-02 (Actual); Study Completion 2015-05-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects reporting local reactions (pain, erythema, and induration) and their severity, as self reported on e-diaries. | 7 days after vaccination
Proportion of subjects reporting systemic events (fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, and new or worsening joint pain) and their severity, as self reported on e-diaries. | 7 days after vaccination

SECONDARY OUTCOMES:
Proportion of subjects in each vaccine group with neutralizing antibody levels (in Neut units/mL) greater than or equal to specified threshold(s). | Up to 12 months post-dose 3
Proportion of subjects in each vaccine group with neutralizing antibody levels, expressed as geometric mean concentrations (GMCs) (in Neut units/mL). | Up to 12 months post-dose 3
Proportion of subjects in each vaccine group with a greater than or equal to 4 and higher fold-rises in neutralizing antibody levels (in Neut units/mL). | Up to 12 months post-dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (6):
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Carolina Phase I Research, LLC, Raleigh, North Carolina
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Clinical Alliance for Research and Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
- Canada (4):
  - Manna Research Inc., Toronto, Ontario
  - Diex Research Montreal Inc, Montreal, Quebec
  - Clinique Medicale St-Louis (recherche) Inc., Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec